CLINICAL TRIAL: NCT01532583
Title: The Outcome of the Transobturator Tape (TOT) Procedure During the Follow-up of 6.5 Years
Brief Title: The Outcome of the Transobturator Tape (TOT) Procedure
Status: Completed | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 13/2005, 15.2.2005
Record Dates: First submitted 2011-11-29; First posted 2012-02-14 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Patients operated on with the TOT
  Interventions: Other: Gynaecological examination, a supine stress test, questionnaires

INTERVENTIONS:
Other: Gynaecological examination, a supine stress test, questionnaires — Gynaecological examination, a supine stress test, questionnaires

SUMMARY:
The aim of our study is to report the subjective and objective outcome of outside-in transobturator technique (TOT) (Monarc®) in long-term follow-up.

This is a follow-up study concerning 191 patients operated on in Turku University Hospital between May 2003 and December 2004 by using TOT. SUI was diagnosed with a positive stress test, the Urinary Incontinence Severity Score (UISS) and the Detrusor Instability Score (DIS). After a mean of 6.5 years evaluation included a gynecological examination and a supine stress test. Subjective outcome was evaluated with UISS, DIS, a visual analogue scale (VAS), a questionnaire of subjective evaluation of continence, EuroQoL-5D, EQ-5D VAS and short versions of IIQ-7 and UDI-6. Objective cure was defined as negative stress test and an absence of reoperation for SUI during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* 191 patients operated on with the TOT procedure between May 2003 and December 2004 at the Department of Obstetrics and Gynecology in the Turku University Hospital.

Exclusion Criteria:

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 191 female patients with genuine or recurrent stress urinary incontinence or mixed incontinence operated on with the TOT procedure at the mean of 6.5 years ago
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2009-01; Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Objective outcome of the TOT operation, which was evaluated with stress test and need for reoperation for urinary incontinence. | 8 years

SECONDARY OUTCOMES:
Subjective outcome of the TOT operation which was assessed with evaluated questionnaires. | 8 years

CONTACTS AND LOCATIONS:
Locations (1):
- Turku university hospital, Turku, Finland